CLINICAL TRIAL: NCT02659735
Title: A Phase 1, Open-label, 2-panel, Randomized, Crossover Study in Healthy Adult Subjects to Assess the Relative Oral Bioavailability of a Single 600-mg Dose of JNJ-63623872 Administered as Oral Concept Formulations Compared to the Current Tablet Formulation, Under Fed and Fasted Conditions
Brief Title: A Study to Assess the Relative Oral Bioavailability of JNJ-63623872 Administered as Oral Concept Formulations Compared to the Current Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108109; 63623872FLZ1006 (Other: Janssen Research & Development, LLC); 2015-002299-26 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Influenza A Virus
Keywords: Influenza A virus; JNJ-63623872; Healthy
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Panel 1: Treatment ADBC (Experimental): Participants will receive Treatment A (600 milligram [mg] JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fed conditions) in Period 1; followed by Treatment D (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #3 [test 3] under fed conditions) in Period 2; followed by Treatment B (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1 [test 1] under fed conditions) in Period 3; followed by Treatment C (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #2 [test 2] under fed conditions) in Period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 1: Treatment BACD (Experimental): Participants will receive Treatment B (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1 [test 1] under fed conditions) in Period 1; followed by Treatment A (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fed conditions) in Period 2; followed by Treatment C (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #2 [test 2] under fed conditions) in Period 3; followed by Treatment D (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #3 [test 3] under fed conditions) in Period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel I: Treatment CBDA (Experimental): Participants will receive Treatment C (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #2 [test 2] under fed conditions) in Period 1; followed by Treatment B (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1 [test 1] under fed conditions) in Period 2; followed by Treatment D (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #3 [test 3] under fed conditions) in Period 3; followed by Treatment A (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fed conditions) in Period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel I: Treatment DCAB (Experimental): Participants will receive Treatment D (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #3 [test 3] under fed conditions) in Period 1; followed by Treatment C (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #2 [test 2] under fed conditions) in Period 2; followed by Treatment A (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fed conditions) in Period 3; followed by Treatment B (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1 [test 1] under fed conditions) in Period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment EFG (Experimental): Participants will receive Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 1; followed by Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 2; followed by Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment FGE (Experimental): Participants will receive Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 1; followed by Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 2; followed by Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment GEF (Experimental): Participants will receive Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 1; followed by Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 2; followed by Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment GFE (Experimental): Participants will receive Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 1; followed by Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 2; followed by Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment FEG (Experimental): Participants will receive Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 1; followed by Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 2; followed by Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg
- Panel 2: Treatment EGF (Experimental): Participants will receive Treatment E (600 mg JNJ-63623872 formulated as the 300 mg oral tablet [reference] under fasted conditions) in Period 1; followed by Treatment G (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 5] under fed conditions) in Period 2; followed by Treatment F (600 mg JNJ-63623872 formulated as the 600 mg oral concept formulation #1, #2 or #3 [test 4] under fasted conditions) in Period 3. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-63623872 300 milligram (mg); Drug: JNJ-63623872 600 mg

INTERVENTIONS:
Drug: JNJ-63623872 300 milligram (mg) — Participants will receive 600 milligram (mg) JNJ-63623872 formulated as the 300 mg oral tablet on Day 1.
Drug: JNJ-63623872 600 mg — Participants will receive 600 mg JNJ-63623872 formulated as 600 mg oral concept formulation #1 on Day 1.
Drug: JNJ-63623872 600 mg — Participants will receive 600 mg JNJ-63623872 formulated as 600 mg oral concept formulation #2 on Day 1.
Drug: JNJ-63623872 600 mg — Participants will receive 600 mg JNJ-63623872 formulated as 600 mg oral concept formulation #3 on Day 1.

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of JNJ-63623872 following administration of a single dose as three different concept formulations with that following administration of the current formulation, under both fed and fasted conditions, in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 2-panel, randomized, crossover study in healthy adult participants to assess the relative bioavailability JNJ-63623872. The study population will consist of 48 healthy adult participants, equally divided over 2 panels: 24 participants in Panel 1 and 24 participants in Panel 2. participants will be randomized within each panel. Participants will not be randomized between panels. Panels 1 and 2 will be performed sequentially. Participants having participated in one panel cannot also participate in the other panel. In Panel 1, during 4 subsequent treatment sessions (Periods I, II, III and IV), each participant will receive 4 treatments (Treatments A, B, C, and D), randomized according to a classical 4 sequence, 4 period Williams design. In Panel 2, during 3 subsequent treatment sessions (Periods I, II and III), each participant will receive 3 treatments (Treatments E, F, and G) randomized according to a classical 6 sequence, 3 period Williams design. Primarily, pharmacokinetic parameters will be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* A female participants must be either: a) Not of childbearing potential: postmenopausal greater than (>) 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 international Unit/Liter (IU/L); OR b) Permanently sterilized (example, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or otherwise incapable of becoming pregnant; OR c) If of childbearing potential and heterosexually active, be practicing an effective method of contraception before entry and agree to continue to use two effective methods of contraception throughout the study and for at least 90 days after receiving the last dose of study drug
* A female participant (except if postmenopausal) must have a negative serum beta human chorionic gonadotropin (beta hCG) pregnancy test at Screening and on Day -1
* Participants must have a Body Mass Index (BMI) between 18.0 and 30.0 kilogram per meter^2 (kg/m^2) (extremes included)
* Participants must have a blood pressure (after the participant is supine for at least 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at Screening
* Participants must be non-smokers for at least 3 months prior to Screening

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a past history of heart arrhythmias (extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participant has taken any disallowed therapies before the planned first intake of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Day 1
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Day 1
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) | Day 1
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) | Day 1
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Baseline up to 10 to 14 days after last study drug administration
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Taste Questionnaire Assessment | Day 1
  Participants will answers a questionnaire on taste of the study drug. The questionnaire consists of 4 parts (sweetness, bitterness, flavour and overall); each parts is scored on 4 points , i.e. none, weak, moderate and strong.
Swallowability Assessment | Day 1
  Swallowability will be assessed on a scale of 1-7; how difficult/easy was it to swallow this tablet. In the scale 0=very difficult and 7=very easy.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium